CLINICAL TRIAL: NCT05285566
Title: A Phase IV Randomized, Single-Blind Trial of Liposomal Bupivacaine (Exparel®) for Pain Control in Costal Cartilage Harvest
Brief Title: Pain Control for Undergoing Costal Cartilage Harvesting
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael D. Olson, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-008473
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Nasal Surgery
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exparel® Injection Group (Experimental): On the day of clinically indicated nasal surgery the surgical wound on the chest, where the rib cartilage is removed, will be injected with Exparel®
  Interventions: Drug: Exparel
- Xylocaine® Injection Group (Active Comparator): On the day of clinically indicated nasal surgery the surgical wound on the chest, where the rib cartilage is removed, will be injected with Xylocaine® as part of standard of care.
  Interventions: Drug: Xylocaine

INTERVENTIONS:
Drug: Exparel — 106mg (8 mL) subcutaneous injection injected after costal cartilage harvest
  Other Names: Liposomal bupivacaine
  Arms: Exparel® Injection Group
Drug: Xylocaine — 8 mL of 1% lidocaine with 1:100,000 of epinephrine into costal cartilage wound site
  Other Names: Lidocaine
  Arms: Xylocaine® Injection Group

SUMMARY:
The purpose of this study is to find out whether injecting the U.S. Food and Drug Administration (FDA) approved drug EXPAREL®, a long acting (approximately 96 hours) numbing medication, will reduce pain after rib cartilage removal in comparison to the standard injection of XYLOCAINE®.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of functional nasal obstruction or aesthetic nasal concern requiring nasal surgery with costal cartilage harvest.
* Willing and able to understand and provide written informed consent.

Exclusion Criteria:

* Known pregnancy.
* Women who are currently nursing a child.
* History of coagulopathy; such as hemophilia or Von Willebrand disease, or any congenital or acquired bleeding disorder.
* Use of anticoagulation medication during the study, i.e. aspirin, Coumadin, Plavix, or medications similar in class to these medications will exclude the patient from participation.
* Inability to provide informed consent (patients under guardianship).
* Known hypersensitivity to local anesthetics
* History of cardiac disease; such as current impaired cardiovascular function, past history of myocardial infarction, congenital heart disease, current cardiac symptoms, i.e. angina, shortness of breath, or chest pain as determined by history or review of the medical record.
* History of complex pulmonary disease; such as uncontrolled asthma, COPD, or interstitial lung disease as determined by history or review of the medical record.

Impaired renal function as documented in the medical record in the last 3 months with a serum creatinine greater than 1.2 mg/dL or glomerular filtration rate < 60 mL/min/BSA as determined by history or review of the medical record.

- History of or current hepatic disease as documented by liver function test abnormality in the last 3 months as determined by history or review of the medical record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Pain Scores | 7-10 days following the last administration of study treatment
  Measured using a visual analog scale 0=no pain and 10=worst possible
Change in oral pain medication | 7-10 days following the last administration of study treatment
  Total oral pain medication usage self-reported in pain medication diary

SECONDARY OUTCOMES:
Adverse Reactions | 7-10 days following the last administration of study treatment
  Total number of adverse reactions reported to the study agent

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Olson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States